CLINICAL TRIAL: NCT00828204
Title: An Open-Label, Multicenter Study to Evaluate the Safe and Effective Use of the Single-Use Autoinjector With an Avonex® Prefilled Syringe in Multiple Sclerosis Subjects
Brief Title: Evaluate the Safe and Effective Use of the Avonex® Single-Use Autoinjector in Multiple Sclerosis Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 108MS302
Record Dates: First submitted 2009-01-20; First posted 2009-01-23 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avonex Single-Use Autoinjector (Experimental): Participants received open label weekly treatment with Avonex 30 mcg intramuscular (IM) injections, provided in Avonex prefilled syringes.
  In the Main Study, injection #1: administration of Avonex prefilled syringe via manual IM injection on Day 1. Injections #2, #3, and #4: administration of Avonex prefilled syringe using the single-use autoinjector on Days 8, 15, and 22, respectively. In the Extension Study, participants were to continue treatment with the Avonex single-use autoinjector for up to an additional 12 weeks.
  Interventions: Device: single-use autoinjector with a prefilled liquid Avonex syringe; Device: Avonex prefilled syringe via manual IM injection; Drug: BG9418 (interferon beta-1a)

INTERVENTIONS:
Device: single-use autoinjector with a prefilled liquid Avonex syringe
Device: Avonex prefilled syringe via manual IM injection
Drug: BG9418 (interferon beta-1a)
  Other Names: Avonex

SUMMARY:
The primary objective of the study was to evaluate the safe and effective use of the single-use autoinjector for the intramuscular (IM) delivery of liquid Avonex® (interferon beta-1a) in participants with multiple sclerosis (MS).

DETAILED DESCRIPTION:
The Main Study was a 4-week treatment period which consisted of 1 Avonex manual injection using a prefilled syringe, followed by 3 Avonex injections using the single-use autoinjector. The Extension Study was designed to provide continuation of treatment with the Avonex single-use autoinjector to eligible participants who completed the Main Study for up to an additional 12 weeks, and to obtain additional safety and preference data for the Avonex single-use autoinjector.

Participants were enrolled under the initial study protocol (Initial Subject Subset); the study was subsequently suspended. Changes were made to the protocol (including modifications to the autoinjector needle), and additional participants were enrolled (Main Subject Subset).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Must be 18 to 65 years old, inclusive, at the time of informed consent.
3. Must currently be self-administering Avonex Prefilled Syringes to treat MS and must have been self-administering Avonex Prefilled Syringes for the 12 weeks prior to the Screening Visit.
4. In the investigator's opinion, subjects must be willing and able to self-administer all injections required by the protocol.
5. Must speak English.
6. All male subjects and female subjects of child-bearing potential must practice effective contraception during the study.

Exclusion Criteria:

1. History of seizure disorder or unexplained blackouts OR history of a seizure within 3 months prior to the Screening Visit.
2. History of suicidal ideation within 3 months prior to Day 1 or an episode of severe depression within 3 months prior to Day 1. Severe depression is defined as any episode of depression that requires hospitalization, or the initiation of antidepressant therapy, or an increase in the dose of an existing regimen of antidepressant therapy. NOTE: Subjects receiving ongoing antidepressant therapy are not excluded from the study unless the dose has been increased within the 3 months prior to the Screening Visit.
3. Clinically significant local infection (for example cellulitis, abscess) or systemic infection (pneumonia, septicemia), at the discretion of the Investigator.
4. Known history of Human Immunodeficiency Virus (HIV).
5. Known history of, or positive test result for hepatitis C virus (test for hepatitis C virus antibody [HCV Ab]) or Hepatitis B virus (test for Hepatitis B Surface Antigen [HBsAg] and/or Hepatitis B Core Antibody [HBcAb]).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (16):
- United States (16):
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Maitland, Florida
  - Research Site, Atlanta, Georgia
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Research Site, Boston, Massachusetts
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - Research Site, Buffalo, New York
  - Comprehensive Multiple Sclerosis Care Center, Patchogue, New York
  - Research Site, Charlotte, North Carolina
  - Neurology & Neuroscience Associates, Inc., Akron, Ohio
  - Research Site, Dallas, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Charleston, West Virginia

REFERENCES:
- [Derived] Phillips JT, Fox E, Grainger W, Tuccillo D, Liu S, Deykin A. An open-label, multicenter study to evaluate the safe and effective use of the single-use autoinjector with an Avonex(R) prefilled syringe in multiple sclerosis subjects. BMC Neurol. 2011 Oct 14;11:126. doi: 10.1186/1471-2377-11-126. PMID 21999176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in the following stages: Main Study (Initial Subset and Main Subset enrolled), and Extension Study. Initial subset participants were withdrawn when the study was suspended. After a protocol amendment, the Main Subset participants were enrolled. Only those in the Main Subset had the option to participate in the Extension Study.
Groups:
- Avonex Single-Use Autoinjector: Initial Subset: Participants received open label weekly treatment with Avonex 30 mcg intramuscular (IM) injections, provided in Avonex prefilled syringes.
  In the Main Study, injection #1: administration of Avonex prefilled syringe via manual IM injection on Day 1. Injections #2, #3, and #4: administration of Avonex prefilled syringe using the single-use autoinjector on Days 8, 15, and 22, respectively. In the Extension Study, participants were to continue treatment with the Avonex single-use autoinjector for up to an additional 12 weeks.
  Initial Subset participants were enrolled in the Main Study prior to study suspension and could not enroll in the Extension Study.
- Avonex Single-Use Autoinjector: Main Subset: Participants received open label weekly treatment with Avonex 30 mcg intramuscular (IM) injections, provided in Avonex prefilled syringes.
  In the Main Study, injection #1: administration of Avonex prefilled syringe via manual IM injection on Day 1. Injections #2, #3, and #4: administration of Avonex prefilled syringe using the single-use autoinjector on Days 8, 15, and 22, respectively. In the Extension Study, participants were to continue treatment with the Avonex single-use autoinjector for up to an additional 12 weeks.
  Main Subset participants were enrolled after study suspension and could enroll in the Extension Study.
Period: Main Study: Prior to Study Suspension
Arm/Group | Avonex Single-Use Autoinjector: Initial Subset | Avonex Single-Use Autoinjector: Main Subset
Started | 21 | 0 (Main Subset was not enrolled until after study suspension (period 2, below).)
Completed Manual Injection | 21 | 0
Continued With Autoinjector Injections | 19 | 0
Completed | 7 | 0
Not Completed | 14 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Subject Was Withdrawn | 2 | 0
Not completed — Study Suspension | 11 | 0
Period: Main Study: After Study Restart
Arm/Group | Avonex Single-Use Autoinjector: Initial Subset | Avonex Single-Use Autoinjector: Main Subset
Started | 0 (Initial Subset participants did not continue after the study was suspended.) | 74 (After a protocol amendment, the Main Subset participants were enrolled.)
Completed Manual Injection | 0 | 74
Continued With Autoinjector Injections | 0 | 72
Completed | 0 | 71
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Noncompliance | 0 | 1
Period: Extension Study
Arm/Group | Avonex Single-Use Autoinjector: Initial Subset | Avonex Single-Use Autoinjector: Main Subset
Started | 0 (Participation in the Extension Study was not offered to Initial Subset after completing Main Study.) | 64 (Participation in Extension Study was optional for Main Subset participants completing Main Study.)
Completed | 0 | 61
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: This table presents the baseline characteristics for both the Initial Subset and Main Subset populations. As represented in the Participant Flow module, these 2 groups participated prior to and after study suspension, respectively; therefore the total column should not be interpreted as cumulative.
Groups:
- Total: Total of all reporting groups
Arm/Group | Avonex Single-Use Autoinjector: Main Subset | Avonex Single-Use Autoinjector: Initial Subset | Total
Number analyzed (Participants) | 74 | 21 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 21 | 93
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 18 | 82
  Male | 10 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in the Main Subset With Overall Success Using the Avonex Single-Use Autoinjector
Description: A trainer/observer documented the participant's ability to self-inject with the Avonex single-use autoinjector and completed an observation form. Overall success in using the device for each participant was defined as no failures occurring in any step (ie, device set-up, self-administration of injection, and capping/disposal of the device) during the participant's use of the single-use Avonex autoinjector.
Time Frame: Day 22
Population: Participants in the Main Subset who received an injection of Avonex prefilled syringe as a manual IM injection, at least 1 injection of Avonex prefilled syringe using the autoinjector, and had a completed Observation Form were included in the analysis. Missing data were not imputed. All analyses are based on observed data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avonex Single-Use Autoinjector: Main Subset
Number analyzed (Participants) | 70
percentage of participants | 89 [81 to 96]

2. Other Pre Specified Outcome: Number of Participants in the Initial Subset Who Were Satisfied With the Avonex Single-Use Autoinjector
Description: Number of participants in the Initial Subset who answered yes to the question "Were you satisfied with this single-use injector?" on the Subject Satisfaction Questionnaire.
Time Frame: Day 23
Population: Participants in the Initial Subset who received at least 1 injection with autoinjector who had a complete Subject Satisfaction Questionnaire.
Measure: Number; unit: participants
Arm/Group | Avonex Single-Use Autoinjector: Initial Subset
Number analyzed (Participants) | 18
participants | 14

3. Other Pre Specified Outcome: Percentage of Participants With No Erythema, Induration, or Tenderness, and Normal Temperature at the Injection Site After Injection With the Avonex Single-use Autoinjector
Description: The clinician/investigator evaluated the injection site for erythema, induration, and tenderness as none, mild, moderate, or severe after the use of the Avonex single-use autoinjector. Temperature at the injection site was evaluated as normal, warm, or hot. Those participants having no erythema, induration, or tenderness, and normal temperature at the injection site after injection are presented.
Time Frame: Day 1, Day 8 through 22 (highest severity reported between Days 8 and 22)
Population: Participants who received at least one injection with the Avonex single-use autoinjector. Missing data were not imputed.
Measure: Number; unit: percentage of participants
Arm/Group | Avonex Single-Use Autoinjector: Main Subset | Avonex Single-Use Autoinjector: Initial Subset
Number analyzed (Participants) | 72 | 19
percentage of participants
  No Erythema | 65 | 95
  No Induration | 86 | 100
  No Tenderness | 90 | 79
  Normal Temperature | 100 | 100

4. Other Pre Specified Outcome: Mean Score for Ease of Use Grading Scale
Description: Participants scored the ease of use of the Avonex manual injector (Day 1) and single-use autoinjector (Days 8, 15, 22) using a scale that ranged from 0 (extremely difficult) to 10 (extremely easy).
Time Frame: Day 1, Day 8, Day 15, Day 22
Population: Participants who received at least one injection with the Avonex Single-use Autoinjector. Missing data were not imputed. n=number of participants who received an injection and had an assessment at the given timepoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Avonex Single-Use Autoinjector: Main Subset | Avonex Single-Use Autoinjector: Initial Subset
Number analyzed (Participants) | 72 | 19
scores on a scale
  Day 1 (Manual Injection) n=72, 19 | 8.1 (2.64) | 7.4 (2.41)
  Day 8 (Autoinjector) n= 72, 18 | 8.9 (1.96) [0 to 10] | 6.8 (3.39)
  Day 15 (Autoinjector) n=71, 16 | 8.7 (2.47) [0 to 10] | 6.7 (3.07)
  Day 22 (Autoinjector) n=70, 7 | 9.3 (1.87) [1 to 10] | 5.9 (3.13)

5. Other Pre Specified Outcome: Percentage of Participants Who Rated the Avonex Single-use Autoinjector Printed and DVD Training Materials as Very Effective
Description: Participants evaluated how effective the printed and DVD instructions were in educating how to use the Avonex single-use autoinjector. Participants could choose one of the following descriptive answers: not effective at all, somewhat ineffective, neutral, somewhat effective, or very effective.
Time Frame: Day 8, Day 15, Day 22
Population: Participants in the Main Subset who received at least one injection with the Avonex Single-use Autoinjector and submitted an assessment form. n=the number of subjects completing the assessment form at the given timepoint. Missing data were not imputed.
Measure: Number; unit: percentage of participants
Arm/Group | Avonex Single-Use Autoinjector: Main Subset
Number analyzed (Participants) | 72
percentage of participants
  Printed instructions, Day 8; n=68 | 93
  DVD, Day 8; n=69 | 88
  Printed instructions, Day 15; n=42 | 90
  DVD, Day 15; n=10 | 90
  Printed instructions, Day 22; n=24 | 92
  DVD, Day 22; n=9 | 89

6. Other Pre Specified Outcome: Mean Score for Initial Subset on Autoinjector Instructions Grading Scale
Description: Participants in the Initial Subset were asked to answer the question "How satisfied are you with the presentation of the autoinjector instructions?" on a rating scale of 0 (extremely dissatisfied) to 10 (extremely satisfied).
Time Frame: Day 8
Population: Participants in the Initial Subset who received at least one injection with the Avonex single-use autoinjector and completed the grading scale.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Avonex Single-Use Autoinjector: Initial Subset
Number analyzed (Participants) | 18
scores on a scale | 9.5 (0.71)

7. Other Pre Specified Outcome: Percentage of Participants Who Indicated No Difficulty With the Injection Procedure of the Manual Injection or the Avonex Single-use Autoinjector
Description: Participants assessed whether they had experienced any difficulty with the procedure in preparing, injecting, removing, and disposing process after each injection with the Avonex single-use autoinjector by answering yes or no to the following question: "Did you have any difficulty with your injection?" The percentage of participants answering no to this question for both the manual injection on Day 1 and the autoinjector on Days 8. 15 and 22 are presented.
Time Frame: Day 1, Day 8, Day 15, Day 22
Population: Participants in the Main Subset who received at least one injection with the Avonex single-use autoinjector and submitted an assessment of injection procedure form. Missing data were not imputed. n=number of participants with assessment at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Avonex Single-Use Autoinjector: Main Subset
Number analyzed (Participants) | 72
percentage of participants
  Day 1 (Manual Injection); n=70 | 89
  Day 8 (Autoinjector); n=71 | 90
  Day 15 (Autoinjector); n=71 | 90
  Day 22 (Autoinjector); n=71 | 90

8. Other Pre Specified Outcome: Percentage of Participants Who Indicated a Preference for the Avonex Single-use Autoinjector Over the Manual Avonex Prefilled Syringe
Description: Participants were asked whether they preferred using the Avonex single-use autoinjector over the manual Avonex prefilled syringe. Preference was defined as participants answering yes to the following question: Do you prefer this single-use autoinjector over the manual injection?
Time Frame: Day 23
Population: Participants who received at least 1 injection with autoinjector and had a complete questionnaire. Missing data were not imputed.
Measure: Number; unit: percentage of participants
Arm/Group | Avonex Single-Use Autoinjector: Main Subset | Avonex Single-Use Autoinjector: Initial Subset
Number analyzed (Participants) | 70 | 18
percentage of participants | 94 | 53

9. Other Pre Specified Outcome: Mean Pain Score After Injection
Description: Participants scored their pain level after the use of the manual prefilled syringe on Day 1 and the Avonex single-use autoinjector on Days 8, 15, and 22 on a scale ranging from 0 (no pain) to 10 (extremely painful).
Time Frame: Day 1, Day 8, Day 15, Day 22
Population: Participants in the Main and Initial Subsets who received at least 1 dose of Avonex injection using the Avonex single-use autoinjector. Missing data were not imputed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Avonex Single-Use Autoinjector: Main Subset | Avonex Single-Use Autoinjector: Initial Subset
Number analyzed (Participants) | 72 | 19
scores on a scale
  Day 1 (Manual Injection) n=72, 19 | 1.7 (1.76) | 2.5 (2.87)
  Day 8 (Autoinjector) n= 72, 18 | 1.0 (1.46) [0 to 7] | 1.9 (2.19)
  Day 15 (Autoinjector) n=71, 16 | 1.3 (1.64) [0 to 6] | 2.1 (1.95)
  Day 22 (Autoinjector) n=70, 7 | 0.7 (1.13) [0 to 6] | 2.4 (2.99)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) treatment-emergent to the autoinjector (from Day 8) through Day 23 (end of Main Study, for the Initial Study Subset), and through Day 107 (end of Extension Period, for the Main Study Subset).
Arm/Group | Avonex Single-Use Autoinjector: Main Subset | Avonex Single-Use Autoinjector: Initial Subset
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/19
Other Adverse Events (participants affected / at risk) | 33/72 | 7/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avonex Single-Use Autoinjector: Main Subset (N=72) | Avonex Single-Use Autoinjector: Initial Subset (N=19)
Acute Sinusitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 1 | 0
Lyme Disease (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0
Bipolar Disorder (Psychiatric disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 1
Multiple Sclerosis Relapse (Nervous system disorders) | 1 | 0
Macular Degeneration (Eye disorders) | 1 | 0
Ulcerative Keratitis (Eye disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Respiratory Tract (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Injection Site Pain (General disorders) | 7 | 4
Injection Site Haematoma (General disorders) | 6 | 1
Influenza Like Illness (General disorders) | 3 | 1
Injection Site Erythema (General disorders) | 3 | 1
Injection Site Haemorrhage (General disorders) | 2 | 0
Injection Site Induration (General disorders) | 2 | 0
Injection Site Pruritus (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Vessel Puncture Site Haematoma (General disorders) | 1 | 0
Vessel Puncture Site Pain (General disorders) | 1 | 0
Body Temperature Increased (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Needle Issue (Injury, poisoning and procedural complications) | 0 | 1

LIMITATIONS AND CAVEATS:
The Initial Subset is too small a population from which to draw conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.